CLINICAL TRIAL: NCT04460365
Title: European Nutrition in Glaucoma Management Trial
Acronym: ENIGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Eye Research Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/378/1535
Record Dates: First submitted 2020-03-02; First posted 2020-07-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma, Open-Angle
Keywords: multisensory integration; macular pigment; lutein; zeaxanthin; meso-zeaxanthin; cognitive function; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Lutein; Zeaxanthins; meso-zeaxanthin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Softgel capsules: 10 mg Lutein, 2 mg zeaxanthin, 10 mg meso-zeaxanthin once a day with a meal for 18 months
  Interventions: Dietary Supplement: 10 mg Lutein, 2 mg zeaxanthin, 10 mg meso-zeaxanthin
- Placebo (Placebo Comparator): Identical capsule containing no active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 10 mg Lutein, 2 mg zeaxanthin, 10 mg meso-zeaxanthin — This is a lutein (10mg), zeaxanthin (2mg) and meso-zeaxanthin (10mg) one-a-day food supplement which combines all three macular carotenoids.
  These three nutrients are found at the back of the eye, at the macula, where they form the macular pigment (yellow colour). Meso-zeaxanthin is particularly concentrated at the centre of this pigment.
  Lutein and zeaxanthin can be found in fruits and dark green leafy vegetables and meso-zeaxanthin is present in some species of fish and seafood.
  Arms: Active
Other: Placebo — Softgel capsule containing sunflower oil (no active ingredients)
  Arms: Placebo

SUMMARY:
European Nutrition in Glaucoma Management (ENIGMA) trial will evaluate the effect of 18-month supplementation with lutein, zeaxanthin and meso-zeaxanthin on macular pigment (MP) levels, vision, cognition and serum biomarkers of inflammation and oxidative stress in glaucoma patients.

This study comprises a randomised, placebo controlled and double masked clinical trial designed to establish MP response to supplementation with lutein, zeaxanthin and meso-zeaxanthin over an 18-month period. The study will also investigate the relationship between macular pigment, cognitive function, oxidative stress and inflammation, and determine the impact of dietary supplementation on vision, retinal structure, quality of life and cognitive function among glaucoma subjects.

DETAILED DESCRIPTION:
This is a research study looking at the effects of dietary MP supplementation in glaucoma patients. Glaucoma can cause irreversible visual impairment. Current treatment modalities only halt disease progression and do not improve visual function. It is important to understand that poor visual function can have major consequences to an individual's day-to-day tasks such as increased risk of falls and automobile accidents.

Disability glare is commonly experienced by eye disease patients, including those with glaucoma, and has been shown to be present even in those who are mildly affected by the disease. MP is a blue-light filter that plays an important role in visual performance including glare sensitivity. Moreover, MP is a potent antioxidant, and it is widely known that oxidative stress is involved in the pathogenesis of glaucoma, both at the level of retinal ganglion cells and trabecular meshwork.

Glaucoma and cognitive decline are both neurodegenerative processes that share several antecedents. The clustering of degenerative disorders towards the end of life is thought to be the result of cumulative and lifelong oxidative injury, and is consistent with the free radical theory of aging. Observational studies have revealed links between the two conditions. The commonalities between glaucoma and cognitive decline, including their shared risk factor profile and pathophysiological pathways, suggest a role for exploring common mechanisms and perhaps even a shared therapeutic approach.

The purpose of this study is to investigate the effects of dietary MP supplementation on MP levels, serum biomarkers of inflammation and oxidative stress, vision, retinal structure and cognition in glaucoma patients.

Study design 64 glaucoma participants Treatment arm: 10 mg Lutein, 2 mg zeaxanthin, 10 mg meso-zeaxanthin - 2/3 Placebo arm: Identical capsule containing no active ingredients - 1/3 Duration of intervention: 18 months

At baseline, all glaucoma participants undergo detailed vision assessments including visual acuity, microperimetry, measurement of macular pigment optical density (MPOD) with dual-wavelength fundus autofluorescence technique, optical coherence tomography scans, contrast sensitivity testing with and without glare, photostress recovery time, pupil reaction assessment, lens fluorescence measurement and fill out vision-related and dietary questionnaires. Patients also undergo detailed cognitive assessment including the flanker task, sound-induced flash illusions task, verbal fluency (FAS and animal fluency tests), SKT (short cognitive assessment) and MMSE (mini-mental state examination) tests which provide measures of reaction time, short-term memory, multisensory integration and attention. A blood sample is also collected for analysis of oxidative stress and inflammatory biomarkers.

After the baseline assessments, glaucoma participants are randomised (2:1) to receive a dietary MP supplementation or placebo for 6 months. Each daily dose of the supplement contains 10mg Lutein, 10mg meso-Zeaxanthin and 2mg Zeaxanthin in a softgel capsule. The intervention consists of a daily oral consumption of one softgel capsule (recommended to be consumed with food) for a period of 18 months, with patients compliance checks and re-supply of supplement every 6 months. The placebo looks identical to the active supplement in its preparation size, colour, smell and taste. It contains no active ingredients.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma patients aged 18 years or older

  1. Primary open-angle glaucoma (POAG)
  2. Normal-tension glaucoma (NTG)
  3. Pseudoexfoliative glaucoma
  4. Pigment dispersion glaucoma
* Best corrected visual acuity of better than 6/12 in the study eye (logMAR <0.3)
* Either gender
* Able to give informed consent, make the required study follow-up visits and adhere to trial protocol

Exclusion Criteria:

* Underlying ocular disease such as age-related macular degeneration, diabetic retinopathy or moderate to significant cataract (patients with established cataract who are likely to progress)
* Best corrected visual acuity of worse than 6/12 in the study eye (logMAR > 0.3)
* History of diabetes mellitus, any type of dementia (e.g. Alzheimer's has been shown to be associated with lower macular pigment levels) or other significant systemic condition that might affect capacity to complete the trial
* MMSE score < 26
* Individuals taking dietary macular pigment supplements (containing lutein, zeaxanthin and meso-zeaxanthin, such as MacuShield, Ocuvite Lutein/Complete, I-Caps etc.) in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Change in MPOD in response to treatment from baseline at 18 months | 18 months
  Change in MPOD measured at each study visit from baseline to 18 months will be evaluated between active and placebo arms

SECONDARY OUTCOMES:
Change in multisensory integration from baseline following 18 months supplementation | 18 months
  Multisensory integration will be assessed using a sound-induced flash illusions task (SIFI). Change in SIFI scores will be assessed between active and placebo treatment arms from baseline to 18 months
Change in flanker task scores (reaction time and attention) from baseline following 18 months supplementation | 18 months
  Change in flanker task scores will be assessed between active and placebo treatment arms from baseline to 18 months
Change in SKT (Syndrom-Kurztest) score from baseline following 18 months supplementation | 18 months
  SKT is a short cognitive battery of tests that evaluates general cognitive function. Change in SKT score will be assessed between active and placebo treatment arms from baseline to 18 months
Change in verbal fluency (FAS score) from baseline following 18 months supplementation | 18 months
  Change in verbal fluency assessed using the FAS test will be evaluated between active and placebo treatment arms from baseline to 18 months
Change in verbal fluency (animal fluency test) from baseline following 18 months supplementation | 18 months
  Change in verbal fluency assessed using the animal fluency test will be evaluated between active and placebo treatment arms from baseline to 18 months
Change in Visual Acuity in response to treatment from baseline at 18 months | 18 months
  Change in Visual Acuity will be evaluated between active and placebo treatment arms from baseline to 18 months
Change in Contrast Sensitivity in response to treatment from baseline at 18 months | 18 months
  Change in Contrast Sensitivity under photopic and mesopic conditions at 1.5, 3, 6, 12 and 18 cycles per degree will be evaluated between active and placebo treatment arms from baseline to 18 months, using the FACT device
Change in incremental light sensitivity in response to treatment from baseline at 18 months | 18 months
  Change in Microperimetry average threshold will be evaluated between active and placebo treatment arms from baseline to 18 months, using the Maia device
Change in Retinal Thickness parameters in response to treatment from baseline at 18 months | 18 months
  Change in Retinal Thickness parameters will be evaluated between active and placebo treatment arms from baseline to 18 months, using the Spectralis OCT device
Change in serum biomarkers of inflammation (C-reactive protein) from baseline following 18 months supplementation | 18 months
  Inflammation will be assessed using the C-reactive protein biomarker measured in serum
Change in serum biomarkers of oxidative stress (Oxidized LDL) from baseline following 18 months supplementation | 18 months
  Oxidative stress will be assessed using the Oxidized LDL biomarker measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: James Loughman, PhD, Principal Investigator — Head of the Centre for Eye Research Ireland, Professor
Locations (1):
- Centre for Eye Research Ireland, Dublin, Co. Dublin, Ireland

REFERENCES:
- [Derived] Loughman J, Loskutova E, Butler JS, Siah WF, O'Brien C. Macular Pigment Response to Lutein, Zeaxanthin, and Meso-zeaxanthin Supplementation in Open-Angle Glaucoma: A Randomized Controlled Trial. Ophthalmol Sci. 2021 Jul 11;1(3):100039. doi: 10.1016/j.xops.2021.100039. eCollection 2021 Sep. PMID 36247822